CLINICAL TRIAL: NCT05125159
Title: Randomized Trial of Angioplasty Guidewire-Assisted Transseptal Puncture Technique Versus Conventional Technique for Left Atrial Access in Left Atrial Appendage Occlusion
Brief Title: Angioplasty Guidewire-Assisted Versus Conventional Transseptal Puncture for Left Atrial Appendage Occlusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AGILE-LA Study
Record Dates: First submitted 2021-10-31; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: 150 patients will be randomized in a 1:1, single-blinded fashion to 1 of 2 transseptal groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- angioplasty guidewire-assisted transseptal group (Experimental): Patients randomized to the angioplasty guidewire-assisted transseptal puncture (GW-TSP) group will undergo transseptal puncture with angioplasty guidewire-assistance.
  Interventions: Procedure: angioplasty guidewire-assisted transseptal puncture or Standard conventional transseptal puncture
- Conventional transseptal group (Sham Comparator): Patients randomized to the conventional transseptal group (Standard Group) will undergo transseptal puncture with BRK needle (St. Jude Medical).
  Interventions: Procedure: angioplasty guidewire-assisted transseptal puncture or Standard conventional transseptal puncture

INTERVENTIONS:
Procedure: angioplasty guidewire-assisted transseptal puncture or Standard conventional transseptal puncture — Patients randomized to the angioplasty guidewire-assisted transseptal puncture (GW-TSP) group will undergo transseptal puncture with angioplasty guidewire-assistance.
  Patients randomized to the conventional transseptal group (Standard Group) will undergo transseptal puncture with BRK needle (St. Jude Medical).

SUMMARY:
This will be a prospective, single-blinded, three-center, randomized, controlled trial comparing the effectiveness and safety of angioplasty guidewire-assisted transseptal puncture (GW-TSP) technique to transseptal left atrial (LA) access with conventional transseptal puncture with standard transseptal equipment (CON-TSP) in patients undergoing left atrial appendage occlusion (LAAO) procedure for atrial fibrillation. The targeted population will consist of patients with atrial fibrillation undergoing LAAO.

DETAILED DESCRIPTION:
Transseptal catheterization is a critical step for left atrial interventions (atrial fibrillation ablation, LA appendage closure, mitral valve interventions). The availability of suitable tools and techniques is essential to safely perform the TSP, effectively deliver radiofrequency lesions, deploy LA devices, and anticipate difficult procedural situations in which complications may arise. Historically, a conventional Brockenbrough (BRK) needle has been used for this procedure to mechanically puncture the fossa ovalis, which has been well described in the literature. Although generally safe, serious complications such as perforation of the atrial wall or aorta can occur.

This study is intended to assess the safety, performance and usability of the angioplasty guidewire in facilitating access to the left atrium during LAAO procedures for the treatment of atrial fibrillation (AF). Moreover, the study will assess the impact of the GW-TSP on procedural times, including time to achieve left atrial accesses, total procedure times, total fluoroscopy time. The study is a prospective, single-blinded, three-center, randomized, controlled trial. Enrolled subjects who meet the study inclusion/exclusion criteria will be evaluated during the LAAO procedures and followed until release from hospital post procedure per institutional standard of care. After 30 days, patient will be contacted by telephone to obtain information on their clinical condition and any adverse events; if necessary, a clinic visit may be performed when required by the physician.

ELIGIBILITY:
Inclusion Criteria:

* Patient is referred to receive a LAAO procedure for atrial fibrillation, requiring transseptal access and LA catheterization
* Patients greater than 18 years of age
* Patient has signed the informed consent form and is willing to participate in the clinical study and data collection

Exclusion Criteria:

* Previous left atrial (LA) ablation or LA surgery
* Active Intracardiac Thrombus
* Pre-existing pulmonary vein stenosis or PV stent
* Pre-existing hemidiaphragmatic paralysis
* Contraindication to anticoagulation or radiocontrast materials
* Cardiac valve prosthesis
* Myocardial infarction, PCI / PTCA, or coronary artery stenting during the 3-month period preceding the consent date
* Cardiac surgery during the three-month interval preceding the consent date
* Significant congenital heart defect (including atrial septal defects or PV abnormalities but not including PFO)
* Significant chronic kidney disease (CKD - eGFR <30 µMol/L)
* Uncontrolled hyperthyroidism
* Cerebral ischemic event (strokes or TIAs) during the six-month interval preceding the consent date
* Pregnancy
* Life expectancy less than one year
* Currently participating or anticipated to participate in any other clinical trial of a drug, device or biologic that has the potential to interfere with the results of this study
* Unwilling or unable to comply fully with study procedures and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Total transseptal puncture time | Intraprocedural assessment (within 24 hours)
  in minutes and seconds. (Total time required for left atrial access)

SECONDARY OUTCOMES:
Time from sheath in superior vena cava to sheath in fossa ovalis | Intraprocedural assessment (measured in seconds)
  The time that sheath slides from superior vena cava to fossa ovalis
Time from needle in fossa ovalis to needle in left atrial | Intraprocedural assessment (measured in seconds)
  The time of sheath needle advancement through the septum and into the left atrial.
Time from needle in left atrial to sheath in left atrial | Intraprocedural assessment (measured in seconds)
  Time of needle advancement through the septum to sheath advancement into the left atrial.
Time from sheath in left atrial to sheath in pulmonary vein | Intraprocedural assessment (measured in seconds)
  The time that sheath enters the pulmonary vein after advancement into the left atrial.
Total fluoroscopy time | in seconds
  Total fluoroscopy time
Total procedural time | in minutes
  Total procedural time
contrast volume | During or immediately after procedure
  contrast used in transseptal puncture
Procedure related complication rate | Acute peri-procedural complications will be defined as occurring within 30 days of LAAO: during or immediately after procedure, up to 1 day after procedure, up to 30 days after procedure
  The proportion of patients sustaining a procedural complication plausibly related to transseptal puncture; events include pericardial effusion, pericardial tamponade, cardiac perforation, air embolism, aortic root puncture

CONTACTS AND LOCATIONS:
Overall Officials: LY Gu, Study Chair — Shanghai Jiao Tong University, School of Medicine, Affiliated Ren Ji HospitalH
Locations (1):
- Shanghai Jiao Tong University, School of Medicine, Affiliated Ren Ji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu F, Xu B, Qiao Z, Cheng F, Zhou Z, Zou Z, Zang M, Ding S, Hong J, Xie Y, Zhou Y, Huang J, Pu J. Angioplasty Guidewire-Assisted vs. Conventional Transseptal Puncture for Left Atrial Appendage Occlusion: a multicentre randomized controlled trial. Europace. 2023 Dec 6;25(12):euad349. doi: 10.1093/europace/euad349. PMID 38011331